CLINICAL TRIAL: NCT01925924
Title: Resin-modified Glass Ionomer or Composite for Orthodontic Bonding? - a Multi-centre, Randomised, Single Blinded Clinical Trial
Brief Title: RMGI v Composite for Orthodontic Bonding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STH14372
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Malocclusion
Keywords: Dental cements; Orthodontic adhesives; Glass ionomer cement; Tooth demineralization
MeSH Terms: conditions — Malocclusion; Tooth Demineralization | interventions — Composite Resins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resin-modified glass ionomer cement (Experimental): Resin-modified glass ionomer cement is used to attach the fixed orthodontic brackets (brace) to the teeth.
  Interventions: Other: Resin-modified glass ionomer cement
- Composite resin (Active Comparator): Composite resin is used to attach fixed orthodontic brackets (brace)to the teeth.
  Interventions: Other: Composite resin

INTERVENTIONS:
Other: Resin-modified glass ionomer cement — This material contains fluoride
  Other Names: Brand name: Fuji Ortho
  Arms: Resin-modified glass ionomer cement
Other: Composite resin — This material does not include fluoride
  Other Names: Brand name: Transbond
  Arms: Composite resin

SUMMARY:
Demineralization during orthodontic (brace) treatment is a common clinical problem leading to unsightly white or brown marks on the teeth. A recent systematic review has shown little evidence that current methods of delivering fluoride are effective at reducing this problem.

Design: A multi-centre randomised single blinded controlled clinical trial will be conducted with two parallel groups.

Setting: The trial patients will be treated by eight named operators on the Specialist List for Orthodontics held by the General Dental Council and who work either within the hospital service or specialist orthodontic practice. The sample size calculation suggests that each operator will need to treat 40 patients in the trial (approx 1 session per week) plus up to 10 familiarisation patients before.

Planned trial interventions: Brackets will be bonded to all teeth in front of the first permanent molars with either a resin-modified glass ionomer cement (Fuji Ortho LC) or a light cured composite control (Transbond). The material to be bonded will be allocated randomly.

Outcome measures: The two main outcome measures will be the difference in demineralization of the anterior teeth before and after treatment assessed from photographs and the number of debonded brackets during treatment.

DETAILED DESCRIPTION:
Demineralization (dental decay) around fixed appliance components has been reported to occur in up to 95% of cases where brackets are bonded with composite resins. Although early lesions appear clinically as opaque white or brown areas, if mineral loss continues cavitation will occur. Following appliance removal, the lesions may regress or disappear but may still present an aesthetic problem more than 5 years after appliance removal. Fluoride is known to inhibit lesion development and to enhance remineralization following treatment. Resin-modified glass ionomer cements, which release and absorb fluoride, may be used for bracket bonding thereby offering the possibility of less demineralization around bonded attachments. In addition, these cements appear to behave as reliably as composite in terms of bracket failure rate recorded but these data are from case series rather than optimally designed randomised clinical trials. A bonding agent that can behave as reliably as composite and minimize unwanted enamel demineralization would be optimal; saving on restorative costs that may be required should cavitation occur. From the patients perspective, subjective assessment of treatment outcome is likely to be enhanced as ugly demineralised enamel white lesions will be eliminated.

ELIGIBILITY:
Inclusion Criteria:

* 11 years of age or older;
* In good general health;
* Brush his/her teeth at least once per day;
* Have canine and incisor teeth fully erupted and of normal form on either side of upper/lower arch;
* Require upper and/or lower pre-adjusted edgewise fixed appliance therapy;
* Have given written informed consent;
* Be willing and able to comply with the trial regime.

Exclusion Criteria:

* Undergoing orthognathic treatment;
* Patients with a cleft of the lip or palate;
* Patients with any heart condition or disease necessitating antibiotic cover;
* Diabetes mellitus; epilepsy; physical or mental handicap;
* Poor periodontal health, including the presence of supragingival calculus/subgingival calculus/periodontal pocketing greater than 3mm;
* Gross or uncontrolled caries;
* Labial demineralisation on a canine or incisor tooth;
* Absent or peg-shaped lateral incisors;
* Palatal canines and /or ectopic unerupted incisors.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of demineralised white lesions on the teeth | Assessed the day the fixed orthodontic appliance is removed
  Demineralisation will be assessed from standardised colour images of the upper and lower incisors and canines taken pre-treatment and immediately post-debond

SECONDARY OUTCOMES:
The incidence of orthodontic bracket failure | Assessed the day the fixed orthodontic appliance is removed
  All first time bond/band failures will be recorded at each treatment visit and dated in each subject's data collection form for subsequent failure rate assessment and survival analyses

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Benson, PhD, Principal Investigator — University of Sheffield
Locations (5):
- Cork Dental Hospital and School, Cork, Ireland
- United Kingdom (4):
  - Hightown Orthodontics, Crewe, Cheshire
  - Inline Orthodontics, Stevenage, Hertfordshire
  - Charles Clifford Dental Hospital, Sheffield, South Yorkshire
  - The Orthodontic Centre, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Undecided
May share if suitably anonymised

REFERENCES:
- [Derived] Benson PE, Alexander-Abt J, Cotter S, Dyer FMV, Fenesha F, Patel A, Campbell C, Crowley N, Millett DT. Resin-modified glass ionomer cement vs composite for orthodontic bonding: A multicenter, single-blind, randomized controlled trial. Am J Orthod Dentofacial Orthop. 2019 Jan;155(1):10-18. doi: 10.1016/j.ajodo.2018.09.005. PMID 30591153